CLINICAL TRIAL: NCT01158131
Title: Diabetes Prevention in Women With a Recent History of Gestational Diabetes Mellitus (GDM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ellen W. Seely, Ellen W. Seely, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009p002118
Record Dates: First submitted 2010-06-28; First posted 2010-07-08 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational diabetes mellitus (GDM) in the most recent pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle Intervention group (Experimental): Participants in this group will take part in the lifestyle intervention.
  Interventions: Behavioral: Balance after Baby Lifestyle Intervention Program
- Post-gestational diabetes mellitus (GDM) Follow-up Group (No Intervention): Participants in this group will not take part in the intervention.

INTERVENTIONS:
Behavioral: Balance after Baby Lifestyle Intervention Program — Participants in this intervention will receive support from a lifestyle coach and gain access to a website with online presentations that contain healthy eating and physical activity educational tips. Weekly phone conversations with the lifestyle coach, as well as logging diet and physical activity will also be required of intervention participants.
  Arms: Lifestyle Intervention group

SUMMARY:
Many studies have shown that women with a history of gestational diabetes mellitus (GDM) have an increased risk of developing diabetes later in life. The purpose of the study is to test whether a web-based lifestyle intervention program adapted from the NIH sponsored Diabetes Prevention Program (DPP), modified specifically for women with a recent history of GDM, incorporating advice about diet and physical activity, delivered in the first 12 months after delivery will help women lose weight, improve overall health, and decrease their risk factors for type 2 diabetes.

DETAILED DESCRIPTION:
The landmark Diabetes Prevention Program (DPP) demonstrated that intensive lifestyle intervention in people with impaired glucose tolerance (IGT) could reduce the incidence of type 2 diabetes (Knowler, Barrett-Connor et al. 2002). These findings were consistent, regardless of ethnicity, age, body mass index (BMI), gender (Knowler, Barrett-Connor et al. 2002). However, the DPP lacks a specific focus on new mothers with a recent history of gestational diabetes despite their documented high risk for developing Type 2 diabetes. Although there are recommendations that all women with gestational diabetes mellitus (GDM) receive postpartum testing for diabetes and type 2 diabetes risk reduction, study findings suggest that women with a recent history of GDM may be unaware of their risk for future diabetes, and also do not take steps to reduce their risks (Kim et al., 2007). The postpartum period is also a time when many changes occur in a woman's life, with competing responsibilities often altering sleep patterns, work schedules, eating patterns, exercise regularity, and time allocation (Walker, 1999; Swan et al., 2007). New mothers may have difficulties engaging in healthy lifestyle programs because of lack of time and energy, and because of competing work and family demands, including child care (Swan, Kilmartin, and Liaw, 2007).

Modeled around the barriers identified in literature and gleaned from the focus groups and informant interviews of the preliminary study (2009p-000042), we have created a lifestyle/behavioral intervention that utilizes a modified DPP.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female with a diagnosis of gestational diabetes mellitus (GDM) by Carpenter-Coustan criteria (see below) in most recent singleton or twin pregnancy (Carpenter & Coustan, 1982)
* Women with a glucose value >200 mg/dL after a 50-g glucose challenge test at >12 weeks' gestation will also be included
* 18-45 years old
* No personal history of Type 1 or 2 diabetes
* Pre-pregnancy body mass index between 18 and 40 kg/m2
* Six weeks postpartum body mass index between 25 and 50 kg/m2
* Capable of providing informed consent

Exclusion Criteria:

* Pre-pregnancy diagnosis of diabetes (type 1, 2, or a secondary form of diabetes)
* Pre-pregnancy body mass index <18 kg/m2 (underweight) or >40 kg/m2 (morbidly obese)
* Current pregnancy
* Six weeks postpartum body mass index <25 kg/m2 or >50 kg/m2
* Excessive alcohol intake defined as >1 beverage per night or past history of alcohol abuse (within the previous 5 years)
* Current or past recreational drug use (within the previous 5 years)
* Diagnosis of diseases associated with glucose metabolism
* Taking certain prescription medication including glucocorticoids, atypical antipsychotics associated with weight gain (such as respirdal(respiradone), clozapine (klozaril), olanzapine (zyprexa), quetiapine (seroquel), etc.) or weight loss medications including prescription, non-prescription or herbal medications
* Personal history of breast cancer or any other type of cancer other than a basal cell skin cancer
* Personal history of cardiovascular disease (coronary artery disease, congestive heart failure, valvular heart disease, stroke, transient ischemic attack, or intermittent claudication), kidney disease, liver disease, venous or arterial thromboembolic disease, adrenal insufficiency, depression requiring hospitalization within the past 6 months, or non-pregnancy related illness requiring overnight hospitalization in the past 6 months
* Underlying disease/treatment that might interfere with participation in/completion of the study (e.g., significant gastrointestinal conditions, major psychiatric disorders, and others at the discretion of the study clinician)
* Other active medical problems detected by examination or laboratory testing
* Plans to be in a different geographic area within the year
* Unable to give informed consent
* Non-English speaking

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2009-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Postpartum weight loss | 12 months after delivery
  Postpartum weight loss for all subjects will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen W Seely, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Nicklas JM, Zera CA, England LJ, Rosner BA, Horton E, Levkoff SE, Seely EW. A web-based lifestyle intervention for women with recent gestational diabetes mellitus: a randomized controlled trial. Obstet Gynecol. 2014 Sep;124(3):563-570. doi: 10.1097/AOG.0000000000000420. PMID 25162257
- [Derived] Nicklas JM, Miller LJ, Zera CA, Davis RB, Levkoff SE, Seely EW. Factors associated with depressive symptoms in the early postpartum period among women with recent gestational diabetes mellitus. Matern Child Health J. 2013 Nov;17(9):1665-72. doi: 10.1007/s10995-012-1180-y. PMID 23124798